CLINICAL TRIAL: NCT05492448
Title: A Randomized Double-Blind Controlled Study Comparing the Effects of Probiotic Adjuvant Therapy on the Improvement of Lung Function and Blood Sugar in Patients With Type 2 Diabetes and Chronic Obstruction Pulmonary Disease
Brief Title: Probiotic on Type 2 Diabetes and Chronic Obstruction Pulmonary Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Glac Biotech Co., Ltd (Industry)
Responsible Party: Principal Investigator, Hsieh-Hsun Ho, R&D Director, Glac Biotech Co., Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMRP12110N
Record Dates: First submitted 2022-08-01; First posted 2022-08-08 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes; Chronic Obstructive Pulmonary Disease
Keywords: Diabetes mellitus; Chronic obstructive pulmonary disease; Gut microbiota; Probiotics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- L. salivarius AP-32 and L. reuteri GL-104 (Experimental)
  Interventions: Dietary Supplement: L. salivarius AP-32 and L. reuteri GL-104
- L. reuteri GL-104 (Experimental)
  Interventions: Dietary Supplement: L. reuteri GL-104

INTERVENTIONS:
Dietary Supplement: Placebo — Subjects take one pack containing maltodextrin twice daily after breakfast and dinner.
  Arms: Placebo
Dietary Supplement: L. salivarius AP-32 and L. reuteri GL-104 — Subjects take one pack containing L. salivarius AP-32 and L. reuteri GL-104 twice daily after breakfast and dinner.
  Arms: L. salivarius AP-32 and L. reuteri GL-104
Dietary Supplement: L. reuteri GL-104 — Subjects take one pack containing L. reuteri GL-104 twice daily after breakfast and dinner.
  Arms: L. reuteri GL-104

SUMMARY:
This trial is a randomized, double-blind, parallel placebo clinical trial, the purpose of which is to investigate whether the adjuvant therapy of using probiotics during the treatment of diabetic patients can decrease blood sugar levels significantly in comparison with placebo, and observe if the reduced lung function could be recovered in patients with type 2 diabetes (T2DM) and chronic obstructive pulmonary disease (COPD) simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are between 50-85 years old, and clinical diagnosis of T2DM (HbA1c ≥ 6.5% or fasting plasma glucose ≥ 126 mg/dL or oral glucose tolerance test 2-hour plasma glucose ≥ 200 mg/dL).
* Patients with stable pulmonary obstruction (pulmonary function FEV1/FVC <0.7) with symptoms of pulmonary obstruction.
* Subjects can cooperate with the collection of experimental specimens and return for regular visits.
* The patient or family members have signed the informed consent form.
* The patient must receive adjuvant treatment with probiotic for 12 weeks.

Exclusion Criteria:

* The patient or caregiver is unable to follow the physician's instructions for the trial, including the completed symptom assessment form and compliance with medication.
* The patient has a history of related allergic reactions, or the use of other highly sensitive or contraindicated drugs (Allergy to antibiotics or antipyretics).
* The patient have taken oral immunosuppressive drugs, intravenous steroids or T cell inhibitor ointments within the past 2 weeks.
* The patient has consumed probiotic-related products (including drops, lozenges, capsules, powder and yogurt) within the past 1 month.
* The patient received high doses of steroids within the past 1 month.
* The patient with active infection or severe pulmonary disease (eg, tuberculosis, bronchiectasis, or fibrosis).
* The patient is receiving treatment for a major disease or congenital disease.
* The patient is not suitable to participate in the trial as assessed by the professional physician.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in concentration of glycated hemoglobin (HbA1c). | Before and after 4-, 12-week intervention.
  Changes in concentration of HbA1c were assessed before and after 4-, 12-week intervention.
Changes in ratio of forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC). | Before and after 4-, 12-week intervention.
  Changes in ratio of FEV1/FVC were assessed by bronchodilator test before and after 4-, 12-week intervention.

SECONDARY OUTCOMES:
Changes in concentration of fasting blood sugar. | Before and after 4-, 12-week intervention.
  Changes in concentration of fasting blood sugar were assessed before and after 4-, 12-week intervention.
Changes in concentration of immune cytokines. | Before and after 4-, 12-week intervention.
  Changes in concentration of immune cytokines were assessed before and after 4-, 12-week intervention.
Changes in scores of modified medical research council (mMRC). | Before and after 4-, 12-week intervention.
  Changes in scores of mMRC were assessed before and after 4-, 12-week intervention. The minimum score is 0 and the maximum score is 4. A higher score means more difficult breathing.
Changes in scores of COPD assessment test (CAT). | Before and after 4-, 12-week intervention.
  Changes in scores of CAT were assessed before and after 4-, 12-week intervention. The minimum score is 0 and the maximum score is 40. A higher score means more seriously affect life.
Changes of the composition in gut microbiota. | Before and after 12-week intervention.
  Changes of the composition in gut microbiota were analyzed by next-generation sequencing (NGS) before and after 12-week intervention.
Changes of the composition in lower respiratory tract microbiota. | Before and after 12-week intervention.
  Changes of the composition in lower respiratory tract microbiota were analyzed by next-generation sequencing (NGS) before and after 12-week intervention.
Changes of concentration in short-chain fatty acid (SCFA) on plasma. | Before and after 12-week intervention.
  Changes of concentration in SCFA on plasma were analyzed by gas chromatography-mass spectrometry before and after 12-week intervention.
Changes of concentration in short-chain fatty acid (SCFA) on stool. | Before and after 12-week intervention.
  Changes of concentration in SCFA on stool were analyzed by gas chromatography-mass spectrometry before and after 12-week intervention.
Changes in scores of modified Bristol stool form scale. | Before and after 4-, 12-week intervention.
  Changes in scores of modified Bristol stool form scale were assessed before and after 4-, 12-week intervention. The questionnaire included the stool form [1 = very hard (small hard lumps), 2 = hard stool (hard sausage shape), 3 = normal stool (sausage to banana shape), 4 = soft stool, 5 = muddy stool, 6 = watery stool], ease of defecation (1 = difficult, 2 = easy, 3 = very easy) and abdominal symptoms [frequency of upper abdominal pain, lower abdominal pain, borborygmus, and flatulence (1 = frequent, 2 = occasional, 3 = almost never)].

CONTACTS AND LOCATIONS:
Locations (1):
- Glac Biotech Co., Ltd., Tainan, Taiwan